CLINICAL TRIAL: NCT01812499
Title: Common Causes of Blood Transfusion Events in a University Hospital: Analysis of Incident Reports.
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S55141
Record Dates: First submitted 2013-02-12; First posted 2013-03-18 (Estimated); Last update posted 2013-03-18 (Estimated); Status verified 2013-02

CONDITIONS: Blood Transfusion Events
Keywords: blood transfusion; adverse event; incident reporting

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Inhospital the blood transfusion process consists of many phases: ordering the blood product, analysis of the blood sample, delivery, transport and storage of the blood product and administration. In each of these phases (near) accidents may occur. A severe transfusion incident refers to the transfusion of a wrong blood product, whereas a near miss is detected before transfusion.

In 2010 the University Hospitals Leuven introduced a new electronic patient incident report system for transfusion events.

In this study the investigators will analyze the reported blood transfusion events to detect the most common causes of blood transfusion events and the weakest link in the blood transfusion chain.

DETAILED DESCRIPTION:
A retrospective survey will be conducted of all transfusion events reported in the University Hospitals Leuven between January 2011 and July 2012. Both severe accidents and near misses will be included.

Data will be drawn from the incident report system. Data concerning the number of transfused blood products will be required from the Medical Administration Service.

Events will be classified according to the severity and the cause of the event. The different settings where the events took place will be compared using a chi-square test (p<0,05).

ELIGIBILITY:
Inclusion Criteria:

* all transfusion events reported in the University Hospitals Leuven between January 2011 and July 2012
* Both severe accidents and near misses were included

Exclusion Criteria:

* Transfusion reactions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients in a university hospital which experienced a transfusion event
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2013-01; Primary Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Severity of inhospital blood transfusion events | up to 1,5 years
  included events will be classified into near misses or severe incidents

SECONDARY OUTCOMES:
Causes of inhospital blood transfusion events | up to 1,5 years
  Events are classified into human error, technical problems, deficiency of the blood product and others.
  Events will also be classified considering the phase in the blood transfusion process.
  Causes will be studied hospital wide and per setting were the event took place.

OTHER OUTCOMES:
Incidence of inhospital blood transfusion events | up to 1,5 years
  The number of transfusion events divided by the total number of transfused blood products in the study period
Is there a relation between misidentification events and the setting where the event took place? | up to 1,5 years
  The different settings where the events took place will be compared using a chi-square test (p<0,05).

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Devos, MD, PhD, Study Director — Department of Hematology, University Hospitals Leuven, Herestraat 49, 3000 Leuven, Belgium; Els Costermans, RN, Principal Investigator — Department of Hematology, University Hospitals Leuven, Herestraat 49, 3000 Leuven, Belgium
Locations (1):
- University Hospitals Leuven, Leuven, Belgium